CLINICAL TRIAL: NCT00903266
Title: Behavioral and Neural Correlates of Melodic-Intonation-Therapy (MIT) and Speech-Repetition-Therapy (SRT) for Patients With Non-fluent Aphasia
Brief Title: Melodic-Intonation-Therapy and Speech-Repetition-Therapy for Patients With Non-fluent Aphasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Gottfried Schlaug, Associate Professor of Neurology; Staff Neurologist, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DC008796; 3R01DC008796-02S1 (NIH); R01DC008796 (NIH)
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Aphasia; Stroke; Cerebrovascular Accident; Apoplexy; Cerebral Infarction
Keywords: Aphasia; Speech Impairment; Stroke; Cerebrovascular Accident; Cerebral Infarction; Brain Ischemia; Brain Infarction; Cerebrovascular Disorder
MeSH Terms: conditions — Aphasia; Stroke; Cerebral Infarction; Speech Disorders; Brain Ischemia; Brain Infarction; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MIT (Experimental): Melodic Intonation Therapy
  Interventions: Behavioral: Melodic Intonation Therapy
- SRT (Active Comparator): Speech-Repetition-Therapy
  Interventions: Behavioral: Speech-Repetition-Therapy
- NTC (No Intervention): No-Therapy Control; Patients in this arm will be re-randomized to the two active arms at the end of the NTC period.

INTERVENTIONS:
Behavioral: Melodic Intonation Therapy — MIT emphasizes the prosody of speech through the use of slow, pitched vocalization (singing).
  Arms: MIT
Behavioral: Speech-Repetition-Therapy — Speech-Reception-Therapy is an equally intensive, alternative verbal treatment method developed for this study.
  Arms: SRT

SUMMARY:
We are doing this clinical trial in order to evaluate two different treatments for non-fluent aphasia: Melodic Intonation Therapy (MIT) and Speech Repetition Therapy (SRT). MIT uses a simple form of singing, while SRT uses intensive repetition of a set of words and phrases. We want to see which intensive form of treatment is more effective in leading to an improvement in speech output compared to a no-therapy control period, and whether either treatment can cause changes in brain activity during speaking and changes in brain structure. We will use a technique known as functional Magnetic Resonance Imaging (fMRI) to measure blood flow changes in the brain and structural MRI that assess brain anatomy and connections between brain regions. We will use fMRI to assess brain activity while a patient speaks, sings, and hums. We will assess changes in brain activity and in brain structure by comparing scans done prior to treatment to scans obtained after treatment and we will also examine changes between treatment groups. We will correlate changes in brain activity and brain structure with changes in language test scores.

DETAILED DESCRIPTION:
One of the few accepted treatments for severe non-fluent aphasia is Melodic Intonation Therapy (MIT). Inspired by the common clinical observation that patients can actually sing the lyrics of a song better than they can speak the same words, MIT emphasizes the prosody of speech through the use of slow, pitched vocalization (singing), and has been shown to lead to significant improvements in propositional speech beyond the actual treatment period. It has been hypothesized that this effect is due to the gradual recruitment of right-hemispheric language regions for normal speech production, and this is further supported by our functional magnetic resonance imaging (fMRI) pilot data. Although the MIT-induced treatment effect has been shown in several small case series, it is not clear whether the effect is due to the intensity of the treatment or to the unique, components of MIT that are not found in other, non-intonation-based interventions. Thus, our overall aim is to test our hypothesis that MIT's rehabilitative effect is achieved by using its melodic and rhythmic elements to engage and/or unmask the predominantly right-hemispheric brain regions capable of supporting expressive language function. In order to test this hypothesis, we have developed an experimental design that includes the randomization of chronic stroke patients with persistent, moderate to severe non-fluent aphasia into three parallel groups receiving 1) 75 sessions of Melodic Intonation Therapy (approximately 15 weeks), 2) 75 sessions of an equally intensive, alternative verbal treatment method developed for this study (Speech Repetition Therapy), or 3) an equal period of No Therapy. All patients will undergo two pre-therapy and two post-therapy behavioral assessments in addition to the pre- and post-therapy fMRI studies and structural MRI studies examining the neural correlates of overtly spoken and sung words and phrases.This design allows us to 1) examine the efficacy of MIT over No Therapy, 2) examine the effects of elements specific to MIT (e.g., melodic intonation and rhythmic tapping) by comparing it to a control intervention (SRT) that is similar in structure and intensity of treatment, 3) compare post-therapy effects with pre-therapy baseline variations, and 4) examine post-treatment maintenance effects. Our primary speech outcome measure will be the number of Correct Information Units (CIU)/min produced during spontaneous speech. Secondary outcome measures include correctly named items on standard picture naming tests, timed automatic speech, and linguistically-based measures of phrase and sentence analysis.

ELIGIBILITY:
Inclusion Criteria:

1. 21-80 years of age
2. first-time ischemic left-hemispheric stroke or cerebrovascular accident
3. at least 12 months out from first ischemic stroke
4. right-handed (prior to stroke)
5. diagnosis of non-fluent or dysfluent aphasia

Exclusion Criteria:

1. older than 80 years of age
2. more than 1 stroke
3. presence of metal or metallic or electronic devices that cannot be exposed to the MRI environment
4. a terminal medical condition; history of major neurological or psychiatric diseases (e.g. epilepsy; meningitis, encephalitis)
5. use of psychoactive drugs/medications such as antidepressants, antipsychotic, stimulants
6. active participation in other stroke recovery trials testing experimental interventions

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2020-05 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Correct Information Units (CIU)/min and CIUs/phrase elicited during spontaneous speech | Baseline (x2), midpoint of therapy, end of therapy, 4 weeks after end of therapy

SECONDARY OUTCOMES:
1) Items named on a standard picture naming test; 2) timed automatic speech; 3) linguistically-based measures of phrase and sentence analysis; 4) functional and structural imaging measures | baseline (x2), midpoint of therapy, end of therapy, 4 weeks after end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Schlaug, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center / Harvard Medical School; Andrea Norton, BM, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center / Harvard Medical School, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ozdemir E, Norton A, Schlaug G. Shared and distinct neural correlates of singing and speaking. Neuroimage. 2006 Nov 1;33(2):628-35. doi: 10.1016/j.neuroimage.2006.07.013. Epub 2006 Sep 7. PMID 16956772
- [Background] Norton A, Zipse L, Marchina S, Schlaug G. Melodic intonation therapy: shared insights on how it is done and why it might help. Ann N Y Acad Sci. 2009 Jul;1169:431-6. doi: 10.1111/j.1749-6632.2009.04859.x. PMID 19673819
- [Result] Schlaug G, Marchina S, Norton A. From Singing to Speaking: Why Singing May Lead to Recovery of Expressive Language Function in Patients with Broca's Aphasia. Music Percept. 2008 Apr 1;25(4):315-323. doi: 10.1525/MP.2008.25.4.315. PMID 21197418
- [Result] Schlaug G, Marchina S, Norton A. Evidence for plasticity in white-matter tracts of patients with chronic Broca's aphasia undergoing intense intonation-based speech therapy. Ann N Y Acad Sci. 2009 Jul;1169:385-94. doi: 10.1111/j.1749-6632.2009.04587.x. PMID 19673813
- See also: Under "projects" we provide details of our aphasia studies and other studies currently going on in our laboratory. — http://www.musicianbrain.com